CLINICAL TRIAL: NCT06695910
Title: Modulation of the Brain Fog Scale by Eicosapentaenoic Acid Monoglycerides (MAG-EPA) in Volunteers Who Reported Suffering From Haze or Mental Fatigue on a Regular Basis. Exploratory Study (NBF-MG01).
Brief Title: Modulation of the Brain Fog Scale by Eicosapentaenoic Acid Monoglycerides (MAG-EPA).
Acronym: NBF-MG01
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Samuel Fortin (Industry)
Collaborators: Institut de recherche clinique du littoral (IRCL) (Unknown)
Responsible Party: Sponsor-Investigator, Samuel Fortin, President, SCF Pharma
Organization: SCF Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NBF-MG01
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Brain Fog; Cognitive Health
MeSH Terms: conditions — Mental Fatigue | interventions — 1-eicosapentaenoylglycerol; Docosahexaenoic Acids; Sunflower Oil

STUDY DESIGN:
Intervention Model Description: The study is divided in two phases. Phase 1: Single arm. 8 subjects treated with MAG-EPA over a period of 56 days followed by a 28 days wash-out period.
  Phase 2: Two arms, placebo controlled, double-blind study. 40 subjects are assigned either to MAG-EPA or Placebo (sunflower oil) and are treated over a 112 days period followed by a 28 days wash-out period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1: Exploratory MAG-EPA treatment group (Experimental): This is a single arm phase of the study. Every subject will receive the experimental treatment (MAG-EPA) at 1,5g/day for a period of 8 weeks.
  Interventions: Dietary Supplement: Monoglyceride Eicosapentaenoic acid (omega-3)
- Phase 2: MAG-EPA treatment group (Experimental): This phase of the study is a parallel design. Subjects will be assigned to experimental treatment (MAG-EPA) by randomization. Every subject in this arm will receive the same treatment at 1,5g/day for a period of 16 weeks.
  Interventions: Dietary Supplement: Monoglyceride Eicosapentaenoic acid (omega-3)
- Phase 2: Placebo group (Placebo Comparator): This phase of the study is a parallel design. Subjects will be assigned to Placebo treatment (sunflower oil) by randomization. Every subject will receive the same treatment at 2,0g/day for a period of 16 weeks.
  Interventions: Other: Sunflower Oil

INTERVENTIONS:
Dietary Supplement: Monoglyceride Eicosapentaenoic acid (omega-3) — 515 mg MAG-EPA + 33 mg MAG-DHA per capsule x 3 capsules daily: 1.5g/day (MAG-EPA). Subjects will be treated over a period of 56 days (or 112 days in phase 2) followed by a wash-out period of 28 days.
  Other Names: MAG-EPA
  Arms: Phase 1: Exploratory MAG-EPA treatment group; Phase 2: MAG-EPA treatment group
Other: Sunflower Oil — 698 mg sunflower oil per capsule x 3 capsules: 2.0g/d sunflower oil (Placebo) Subjects will be treated over a period of 112 days followed by a wash-out period of 28 days.
  Other Names: Placebo
  Arms: Phase 2: Placebo group

SUMMARY:
A growing body of studies shows that omega-3s act directly in molecular signaling pathways that reduce inflammation and are thought to have a positive effect on cognitive health. Brain fog is a term that has been popularized in the medical world in the wake of the COVID-19 pandemic. A significant proportion of patients with long COVID reported having cognitive sequelae that were like fogginess. It is defined as a cognitive impairment with characteristic symptoms including problems with concentration, attention and memory, confusion, difficulty understanding what others are saying, reduced mental acuity and mental fatigue. These are episodes of reduced cognitive capacity that are not representative of the person's normal state. This condition can be caused by various factors such as stress, lack of sleep, overwork, depression, hormonal changes due to pregnancy or menopause in women, head injuries, migraine, certain diseases or viral infections, certain medications as well as substance abuse (alcohol and/or street drugs). In this study, we want to test whether omega-3 monoglycerides (MAG-EPA) can modulate the cognitive health of people with brain fog.

DETAILED DESCRIPTION:
The study is divided into two phases. The first will include eight (8) subjects and all will receive the study treatment (MAG-EPA). This is a single arm phase. If signs of improvement in cognitive health are perceived in Phase 1, the study may continue with Phase 2.

Phase two will include forty (40) participants divided into two treatment groups. Assignment to any of the treatment groups will be done by randomization. This phase will be double-blind and controlled by placebo.

Participants will be asked to complete a Brain Fog Scale (BFS) questionnaire at Visit 0, immediately after signing the informed consent form. This questionnaire covers the 14 days preceding Visit 0. The subject will be asked to complete the BFS again at Visit 1, which should take place 14 days after Visit 0. These two questionnaires will provide a self-declared state of the participant's cognitive health in the 28 days preceding the start of treatment. The results of the first two questionnaires (BFS1 and BFS2) will determine whether the participant's cognitive state is severe enough to be eligible for participation in the study. Indeed, an exclusion criterion was written in the protocol to avoid including participants with normal cognitive health. Once enrolled in the study, subjects will be required to complete a BFS every 14 days until day 140, that is to say at each visit as well as at each telephone follow-up in between visits (V1, day 0; T1, day 14; V2, day 28; T2, day 42; V3, day 56; T3, day 70; V4, day 84; T4, day98; V5, day 112; T5, day 126 and V6, day 140).

Treatment will be given to each subject, MAG-EPA in phase 1 or either MAG-EPA or placebo (sunflower oil) in phase 2, to be taken daily from day 0 to day 112 (112 consecutive days in total, also corresponding to 16 weeks of treatment). Every subject will take 3 gelcaps daily for a total dose of 1.5g/day of MAG-EPA or 2.0g/day of sunflower oil. A wash-out period of 28 days, form day 112 to day 140, will follow treatment.

For research purposes, the Omega-3 Index will be measured from blood samples collected at Visit 1, 3, 5 and 6. The Omega-3 Index is a quantitative analysis that measures the blood level of Omega-3. This test is used both to confirm the adherence of subjects to treatment (for all subjects in Phase 1 as well as for the test group in Phase 2) and to control the restriction of Omega-3 in subjects in the control group (the placebo treatment in Phase 2). The Omega-3 Index results are indicative of the treatment received for each subject, therefore, the analysis reports will not be given to research staff who are blinded.

Demographic information will also be noted for every subject to better characterise the study population in each group.

Any adverse change to subject's health will be noted and followed until resolution or other final outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Participant between 19 and 55 years of age.
2. Participant who reports having mental fatigue and/or frequent memory loss and/or difficulty concentrating and/or inattention, confusion and/or a feeling of decreased cognitive acuity for at least 28 days at the time of selection.
3. Participant who obtains a mean score on the BFS screening questionnaires (BFS1 and BFS2) total of at least 30 and/OR who obtains the following minimum score on at least one of the three factors: Factor 1 of at least 15 and/or Factor 2 of at least 15 and/or Factor 3 of at least 12.
4. Available for the entire duration of the study and willing to participate based on the information provided in the ICF duly read and signed by the latter.
5. Absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements, ability to cooperate adequately, ability to understand and observe the instructions of the research staff.
6. Participant having no difficulty in swallowing tablets, capsules or gelcaps.

Exclusion Criteria:

1. Known allergy or intolerance to fish or history of allergic reactions attributable to fish, or to a compound similar to fish oil.
2. Participant who has used omega-3 supplements in the 30 days preceding day 1 of the study.
3. Pregnant or breastfeeding woman as declared by the latter.
4. Presence of dependence on drugs of abuse or alcohol (˃ 3 units of alcohol per day, acute or chronic excessive consumption).
5. Participant included in another clinical study and who is receiving an investigational product or other research treatment.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive health assessment with the Brain Fog Scale (BFS) | Phase 1: Every two (2) weeks over a period of fourteen (14) weeks in total.Phase 2: Every two (2) weeks over a period of twenty-two (22) weeks in total.
  * Evaluate the brain fog of all subjects using the Brain Fog Scale (BFS) before the start of treatment, then every 14 days over a period of 98 days (BFS 1 to 8) in phase 1 or a period of 154 days in phase 2 (BFS 1 to 12).
  * For each BFS measured after the start of treatment (BFS 3 to 8 in phase 1 or BFS 3 to 12 in phase 2), compare the score of each individual factor (Factor 1: mental fatigue; Factor 2: impaired cognitive acuity; Factor 3: confusion) with that obtained at the pre-treatment BFS measures (BFS 1 and 2).
  * For each BFS measured after the start of treatment (BFS 3 to 8 in phase 1 or BFS 3 to 12 in phase 2), compare the total score with that obtained at the pre-treatment BFS measures (BFS 1 and 2).

SECONDARY OUTCOMES:
Omega-3 intake assessment by Omega-3 index analysis | At 0, 4, 8 and 12 weeks in phase 1; At 0, 8, 16 and 20 weeks after the start of the study in Phase 2.
  Measure the subjects' omega-3 index four times during the study (Day 0, Day 28, Day 56 and Day 84 in Phase 1; Day 0, Day 56, Day 112 and Day 140 in Phase 2) to validate if the level of omega-3 index correlates with BFS scores and that the subjects in the test group adhere to the treatment. This measurement is also used to check that subjects in the placebo group are not supplemented with omega-3 during the study. Blinded personnel and subjects will not have access to the results of omega-3 index testing.
Demographic data analysis | From week 0 to 12 in Phase 1; From week 0 to 20 in Phase 2.
  Demographic data such as age, gender, body mass index (BMI), substance use habits (alcohol, tobacco), sports habits, sleep habits as well as daily time spent using electronics will be collected to draw a detailed portrait of the studied population. These data will allow to correct for potential confounding variables in the event of an imbalance between the groups.
Adverse Event reporting | From week 2 to 12 in Phase 1; From week 2 to week 20 in Phase 2.
  Evaluate adverse events potentially related to MAG-EPA throughout the supplementation period as well as during the withdrawal period.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Institut de recherche clinique du littoral (IRCL), Maria, Quebec
  - Institut de recherche clinique du littoral (IRCL), Rimouski, Quebec

IPD SHARING:
Plan to Share IPD: No
Sharing participant data require subject consent for sharing. We do not plan to recontact study subjects for data sharing consent.

REFERENCES:
- [Background] Agata Debowska, Daniel Boduszek, Marek Ochman, Tomasz Hrapkowicz, Martyna Gaweda, Anastazja Pondel, Beata Horeczy, Brain Fog Scale (BFS): Scale development and validation, Personality and Individual Differences Volume 216, 2024, 112427, ISSN 0191-8869.